CLINICAL TRIAL: NCT01099878
Title: Institutional Review Board of Chung Shan Medical University Hospital
Brief Title: Cycling Exercise With Functional Electrical Stimulation Improves Postural Control in Stroke Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Chun-Yu Yeh, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CS07136
Record Dates: First submitted 2010-04-06; First posted 2010-04-08 (Estimated); Last update posted 2010-04-08 (Estimated); Status verified 2010-04

CONDITIONS: Postural Control
Keywords: Cycling Exercise; Functional Electrical Stimulation; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cycling Exercise with Functional Electrical Stimulation (Active Comparator): Cycling Exercise with Functional Electrical Stimulation
  Interventions: Device: Cycling Exercise with Functional Electrical Stimulation
- Cycling Exercise (Placebo Comparator): Cycling Exercise
  Interventions: Device: cycling exercise

INTERVENTIONS:
Device: Cycling Exercise with Functional Electrical Stimulation — The subjects were randomly assigned to the cycling group (CG) performing cycling training without electrical stimulation or the FES-cycling group (FES-CG) performing the same training with the assistance of electrical stimulation. The duration of the training program was 20 minutes. The target cycling cadence was set at 45 rpm.
  Arms: Cycling Exercise with Functional Electrical Stimulation
Device: cycling exercise — The subjects were randomly assigned to the cycling group (CG) performing cycling training without electrical stimulation or the FES-cycling group (FES-CG) performing the same training with the assistance of electrical stimulation. The duration of the training program was 20 minutes. The target cycling cadence was set at 45 rpm.
  Arms: Cycling Exercise

SUMMARY:
The aim of this study is to determine whether a short-term of FES assisted cycling in stroke patients can reduce the muscle tone of the affected leg immediately and the influence the postural control of the subjects.

DETAILED DESCRIPTION:
Patients with stroke frequently results in secondary complications of the neuromuscular system. For post-stroke patients, varying deficits in sensation, muscle strength, muscle tone and associated reaction in the paretic limbs often affect the activities of daily living. Cycling exercise is commonly suggested to improve cardiovascular fitness and functional mobility in patients with stroke. (Janssen, 2008; Holt, 2001; Potempa 1995) Cycling exercise requires less balance capacity and exercise intensity can be controlled. The kinematic patterns of cycling are very similar to that of walking that is one of the most important motor functions to recover in a stroke patient (Ferrante, 2008). Others studies have reported that repetitive passive movement of spastic muscle can increase range motion and reduce stiffness of hypertonic joints in stroke patients (Bressel, 2002; Yeh, 2007). Above studies (Bressel, 2002; Yeh, 2007) suggest leg cyclic movement may be a possible therapeutic modality to reduce hypertonia that is one of the factors disturbed the functional activities for stroke patients.

The application of functional electrical stimulation (FES) is usually used in physical therapy to assist the paretic limb to perform functional tasks (5-7). The previous studies reported the functional tasks of hemiplegic hands are improved after electrical stimulation treatment (Wu, 2006; Santos, 2006). FES has also been used to improve the walking ability of subjects with stroke (Bogataj, 1989; Yan, 2005; Salm, 2006). Clinical studies on central motor neuroplasticity also support the role of goal-oriented, repetitive, active movement in the therapy of paretic limbs to enhance motor recovery and relearning in stroke patients. (Ferrante, 2008) In the first half of the 1980s, FES was applied during cycling exercise on the paretic legs of people with spinal cord injury (SCI). The beneficial effects of cycling exercise via FES have evidenced increases in muscle strength and endurance, increases in bone density, suppression of spasticity, improvement of cardiopulmonary function, and many other physiological and psychological effects of benefit for SCI patients (Donaldson et al., 2000; Gfohler and Lugner, 2000; Gfohler et al., 2001). Recently, similar FES assisted cycling devices have also been used for stroke patients (Janssen, 2008; Ferrante, 2008). They reported that FES assisted training provided increased aerobic capacity and functional performance for them. However, in one study (Janssen, 2008) the functional performance was evaluated by clinical scales which do not reflect the changes on the affected limb influenced by the training exercise. It is worthwhile to realize the effects on the affected leg and the changes on postural control after the FES-cycling training.

A new FES-cycling device (Figure.1), modified from our previous prototype (Chen, 2004), was used in this study. This device combines FES with a cycling system equipped with ankle-foot orthoses. The FES stimulates the quadriceps and hamstring when the affected leg sweeps past a specific angle. The aims of this study were to determine whether a short-term of FES-cycling program in stroke patients can reduce the muscle tone of the affected leg immediately and influence the postural control of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* (1)First-ever stroke with unilateral hemiplegia (Brunnstrom stage ≥3);
* (2)Hypertonia in the paretic leg, modified Ashworth scale (MAS) grade of ≥1;
* (3)Ability to understand and follow verbal commands;

Exclusion Criteria:

* (1)Severe perceptual, cognitive, or sensory deficits;
* (2)History of osteoarthritis, severe cardiopulmonary disease, or vascular disease in the lower limbs;
* (3)Fixed contracture in the paretic lower limb.

Ages: 29 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chun -Yu Yeh, PT, PhD, Principal Investigator — Chung Shan Medical University; Chun-Yu Yeh, PT;PhD, Study Chair — Chung Shan Medical University
Locations (2):
- Taiwan (2):
  - Chun-Yu Yeh, Taichung
  - Chung Shan Medical University, Taichung